CLINICAL TRIAL: NCT03835104
Title: Urine and CRP Tests at the Point-of-care for the Diagnostic Assessment of Acutely Ill Children: a Diagnostic and Prognostic Study
Brief Title: ERNIE4: Urine and CRP Point-of-care Test in Acutely Ill Children
Acronym: ERNIE4
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Covid pandemic caused recruitment to stop
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Ann Van den Bruel, Associate Professor, KU Leuven
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: S61991
Record Dates: First submitted 2019-01-29; First posted 2019-02-08 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Infection
Keywords: diagnosis; sensitivity and specificity; serious infections
MeSH Terms: conditions — Infections; Disease; Hypersensitivity

STUDY DESIGN:
Intervention Model Description: The study is a cluster randomized controlled trial. The general practice is the unit of cluster.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRP in all (Active Comparator): All children will undergo a CRP point-of-care test using a fingerprick of blood and producing a result within 4 minutes using the Afinion 2 (Abbott).
  There will be only 1 test at study entry
  Interventions: Device: CRP point-of-care testing
- CRP in high risk children only (Experimental): Children who are positive on a clinical prediction rule for serious infections in children will undergo CRP point-of-care test using a fingerprick of blood and producing a result within 4 minutes using the Afinion 2 (Abbott).
  There will be only 1 test at study entry
  Interventions: Device: CRP point-of-care testing

INTERVENTIONS:
Device: CRP point-of-care testing — CRP point-of-care test using a fingerprick of blood and producing a result within 4 minutes, using the Afinion 2 (Abbott)

SUMMARY:
This study aims to assess the accuracy of a novel urine test for diagnosing urinary tract infections in acutely ill children presenting to ambulatory care. The accuracy of this novel test will be compared to the accuracy of conventional dipstick testing. In addition, the evidence on urine tests will be added to the existing algorithm for diagnosing serious infections in children. Finally, the study aims to describe the relation between the CRP level at study entry and the duration of symptoms and final diagnosis over the following 30 days.

DETAILED DESCRIPTION:
The design is a cross-sectional cohort study with a nested longitudinal follow-up in acutely children presenting to ambulatory care.

The cross-sectional cohort study will compare an innovative urine test with conventional dipstick testing to establish their relative accuracy to diagnose urinary tract infections, and construct an algorithm consisting of clinical features, urine test results and CRP point-of-care testing to identify serious infections. The longitudinal follow-up study will describe illness trajectories of children with an intermediate CRP test result (5-80 mg/L) at first contact.

The study will run in general practices and community paediatrics in Flanders. Recruitment to the study is expected to last 18 months, with each patient entering the study only once. Children and their parents/guardians will be approached for possible participation in the study by practice staff. There is only one study visit.

Those who agree to participation via written informed consent will have demographics and clinical features recorded. All children will be asked to provide a urine sample on study entry. Subsequently, CRP point-of-care testing will be conducted in all children testing positive on a clinical prediction rule, and in a random sample of children testing negative on that rule. Follow-up information for all children will be collected using general practice notes, hospital records and direct patient/parent contact.

Treatment and other management decisions will be left to the treating physicians' discretion.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 months to 18 years
* Presenting to a general practice or community paediatrics
* Acute illness of a maximum of 10 days
* Parent or guardian is willing and able to give informed consent for participation

Exclusion Criteria:

* Clinically unstable warranting immediate care
* Urinary catheter in situ
* Immunosuppressant medication taken in the previous 30 days
* Trauma is the main presenting problem
* Antibiotics taken in the previous 7 days
* Children who present to community paediatrics as a result of direct GP referral

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 868 (Actual)
Dates: Start 2019-02-12 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-05-22 (Actual)

PRIMARY OUTCOMES:
Urinary tract infection | 3 days
  The number of children with a urinary tract infection based on urine culture

SECONDARY OUTCOMES:
Serious infections | 30 days
  The number of children admitted to hospital for a serious infection which can be pneumonia, sepsis, meningitis, pyelonephritis, osteomyelitis or appendicitis

OTHER OUTCOMES:
Final diagnosis | 30 days
  For children not admitted to hospital, the final diagnosis based on all available clinical information from ambulatory care assessment over 30 days after the index date.
Duration of symptoms | 30 days
  For all children, the duration of symptoms after the index date based on patient diaries
Healthcare resource use | 30 days
  For all children, re-consultation rates in ambulatory care after the index date
Healthcare resource use | 30 days
  For all children, ED attendance after the index date
Healthcare resource use | 30 days
  For all children, hospital admission after the index date

CONTACTS AND LOCATIONS:
Overall Officials: Ann Van den Bruel, MD PhD, Principal Investigator — ACHG, KU Leuven
Locations (1):
- KU Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
Any invitations for data sharing will be assessed on scientific validity, after which a decision will be taken.

REFERENCES:
- [Derived] Boon HA, De Burghgraeve T, Verbakel JY, Van den Bruel A. Point-of-care tests for pediatric urinary tract infections in general practice: a diagnostic accuracy study. Fam Pract. 2022 Jul 19;39(4):616-622. doi: 10.1093/fampra/cmab118. PMID 34633441